CLINICAL TRIAL: NCT00630058
Title: A Phase I, Open-Label, Two-Arm Study of MP-424 in Combination With Peginterferon Alfa 2b and Ribavirin in Patients With Genotype 1b Hepatitis C
Brief Title: A Phase 1 Study of MP-424, Peginterferon Alfa 2b, and Ribavirin in Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: G060-A5
Record Dates: First submitted 2008-02-24; First posted 2008-03-06 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Protease Inhibitor; Telaprevir
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (MP-424 High) (Experimental)
  Interventions: Drug: MP-424(H), PEG-IFN-a-2b, RBV
- Group B (MP-424 Low) (Experimental)
  Interventions: Drug: MP-424 (L), PEG-IFN-a-2b, RBV

INTERVENTIONS:
Drug: MP-424(H), PEG-IFN-a-2b, RBV — MP-424 (three tablets of 250mg tablet at a time, every 8 hours) + PEG-IFN-a-2b + RBV for 12 weeks
  Other Names: Telaprevir
  Arms: Group A (MP-424 High)
Drug: MP-424 (L), PEG-IFN-a-2b, RBV — MP-424 (two tablets of 250mg tablet at a time, every 8 hours) + PEG-IFN-a-2b + RBV for 12 weeks
  Other Names: Telaprevir
  Arms: Group B (MP-424 Low)

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics, HCV RNA kinetics, and other viral characteristics after administration of two arms of MP-424 in combination with Peginterferon Alfa 2b (PEG-IFN-a-2b) and Ribavirin (RBV) to patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with genotype 1b chronic hepatitis C

Exclusion Criteria:

* Patients diagnosed with decompensated cirrhosis
* Patients diagnosed with positive HBs antigen in the test

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumitaka Suzuki, MD, Principal Investigator — Department of Hepatology, Toranomon Hospital
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Suzuki F, Suzuki Y, Sezaki H, Akuta N, Seko Y, Kawamura Y, Hosaka T, Kobayashi M, Saito S, Arase Y, Ikeda K, Mineta R, Watahiki S, Kobayashi M, Nakayasu Y, Tsuda H, Aoki K, Yamada I, Kumada H. Exploratory study on telaprevir given every 8 h at 500 mg or 750 mg with peginterferon-alpha-2b and ribavirin in hepatitis C patients. Hepatol Res. 2013 Jul;43(7):691-701. doi: 10.1111/hepr.12009. Epub 2012 Nov 29. PMID 23190247

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (MP-424 High): Drug: MP-424 750 mg every 8 hours for 12 weeks Other Name: Telaprevir
  Drug: Ribavirin 600 - 1000 mg/day based on body weight for 12 weeks
  Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week for 12 weeks
- Group B (MP-424 Low): Drug: MP-424 500 mg every 8 hours for 12 weeks Other Name: Telaprevir
  Drug: Ribavirin 600 - 1000 mg/day based on body weight for 12 weeks
  Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week for 12 weeks
Period: Overall Study
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Started | 10 | 10
Completed | 6 | 6
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — stopping criteria | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (6.8) | 54.3 (8.5) | 52.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration in Plasma) of MP-424
Description: Data were collected before the first dose in the morning, and at 1, 2.5, 4, 6, 8, 12, 16 and 24 h after the first dose on days 1, 14 and 85.
  Data as pre-dose were collected at Day3, Day8, Day29, Day43 and Day57.
Time Frame: Data were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
μg/mL
  Day 1 (Group A,B:10 cases) | 1.62 (0.43) | 1.45 (0.83)
  Day 14 (Group A,B:10 cases) | 3.96 (1.10) | 3.06 (0.90)
  Day 85 (Group A: 6 cases, Group B: 7 cases) | 3.67 (0.87) | 3.16 (1.10)

2. Primary Outcome: Tmax (Time of Maximum Concentration in Plasma) of MP-424
Description: as for outcome 1
Time Frame: Data were collected at Day1 to Day85
Measure: Median (Full Range); unit: hours
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
hours
  Day 1 (Group A, B:10 cases) | 2.51 [2.25 to 6.00] | 2.54 [2.33 to 8.02]
  Day 14 (Group A, B:10 cases) | 2.50 [2.42 to 5.75] | 2.45 [2.33 to 6.00]
  Day 85 (Group A: 6 cases, Group B: 7 cases) | 3.24 [2.35 to 7.75] | 2.43 [2.33 to 4.00]

3. Primary Outcome: AUC 0-8h (Area Under the Concentration-time Curve From Time Zero to 8 Hours) of MP-424
Description: as for outcome 1
Time Frame: Data were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
μg/mL
  Day 1 (Group A, B: 10 cases) | 7.53 (1.93) | 6.55 (3.73)
  Day 14 (Group A: 9 cases, Group B: 10 cases) | 26.00 (6.77) | 19.94 (5.97)
  Day 85 (Group A: 6 cases, Group B: 7 cases) | 25.00 (5.23) | 21.35 (6.88)

4. Primary Outcome: Ctrough (Minimum Observed Concentration in Plasma) of MP-424
Description: as for outcome 1
Time Frame: Data were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
μg/mL
  Day1 (Group A,B: 10 cases) | 0.846 (0.500) | 0.681 (0.412)
  Day14 (Group A: 9 cases, Group B:10cases) | 2.639 (0.556) | 1.914 (0.717)
  Day85 (Group A: 6 cases, Group B:7cases) | 2.679 (0.355) | 2.105 (0.819)

5. Primary Outcome: T1/2(Time of Half-Life) of MP-424
Description: as for outcome 1
Time Frame: Data were collected at Day1 to Day85
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
hours
  Day1 (Group A: 7 cases, Group B: 8 cases) | 4.87 (2.12) | 4.03 (1.63)
  Day14 (Group A: 8 cases, Group B: 9 cases) | 9.99 (4.37) | 10.00 (6.97)
  Day85 (Group A: 6 cases, Group B: 7 cases) | 9.06 (3.98) | 6.22 (3.64)

6. Secondary Outcome: Antiviral Effects of TVR on HCV Were Assessed by Measuring Plasma HCV RNA Levels
Description: HCV RNA concentrations were determined using the COBAS TaqMan HCV test (Roche Diagnostics). The linear dynamic range of the assay was 1.2-7.8 log10 IU/mL.
Time Frame: 37 weeks
Measure: Mean (Standard Deviation); unit: Log IU / mL
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Number analyzed (Participants) | 10 | 10
Log IU / mL
  Day 1_2.5h (Group A,B: 10 cases) | -0.190 (0.235) | -0.220 (0.329)
  Day 1_4h (Group A,B: 10 cases) | -0.420 (0.264) | -0.390 (0.378)
  Day 1_8h (Group A,B: 10 cases) | -1.300 (0.294) | -1.310 (0.309)
  Day 1_16h (Group A,B: 10 cases) | -2.350 (0.458) | -2.480 (0.286)
  Day 2 (Group A,B: 10 cases) | -3.010 (0.340) | -3.180 (0.220)
  Day 3 (Group A,B: 10 cases) | -3.610 (0.453) | -3.790 (0.407)
  Day 8 (Group A,B: 10 cases) | -4.840 (0.622) | -5.010 (0.551)
  Day 14 (Group A,B: 10 cases) | -5.570 (0.579) | -5.800 (0.554)
  Day 29 (Group A: 10 cases, Group B: 9 cases) | -5.860 (0.611) | -5.978 (0.519)
  Day 43 (Group A: 8 cases, Group B: 8 cases) | -6.000 (0.573) | -5.994 (0.590)
  Day 57 (Group A: 7 cases, Group B: 8 cases) | -5.986 (0.538) | -5.994 (0.539)
  Day 86 (Group A: 6 cases, Group B: 7 cases) | -6.000 (0.588) | -6.114 (0.609)
  Day 92 (Group A: 6 cases, Group B: 7 cases) | -6.000 (0.588) | -6.114 (0.609)
  Day 99 (Group A: 6 cases, Group B: 7 cases) | -6.000 (0.588) | -5.471 (1.065)
  Day 113 (Group A: 6 cases, Group B: 7 cases) | -5.917 (0.564) | -3.457 (2.591)
  Day 141 (Group A: 6 cases, Group B: 7 cases) | -4.233 (2.455) | -3.000 (2.865)
  Day 169 (Group A: 6 cases, Group B: 6 cases) | -3.100 (2.827) | -3.267 (3.067)
  Day 197 (Group A: 6 cases, Group B: 6 cases) | -2.850 (2.947) | -3.283 (3.031)
  Day 225 (Group A: 6 cases, Group B: 6 cases) | -2.633 (2.748) | -3.183 (3.140)
  Day 253 (Group A: 6 cases, Group B: 6 cases) | -1.883 (3.177) | -3.100 (3.234)

ADVERSE EVENTS:
Arm/Group | Group A (MP-424 High) | Group B (MP-424 Low)
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (MP-424 High) (N=10) | Group B (MP-424 Low) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Appetite disorders (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (MP-424 High) (N=10) | Group B (MP-424 Low) (N=10)
Nasopharyngitis (Infections and infestations) | 3 | 4
Anaemia (Blood and lymphatic system disorders) | 9 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 7
Dysgeusia (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 0 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 5
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 8
Malaise (General disorders) | 6 | 5
Influenza like illness (General disorders) | 4 | 2
Low density lipoprotein increased (Investigations) | 0 | 3
Blood uric acid increased (Investigations) | 4 | 4
Blood triglycerides increased (Investigations) | 6 | 5
Blood creatinine increased (Investigations) | 5 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 7
Blood luteinising hormone increased (Investigations) | 1 | 2
Eosinophil percentage increased (Investigations) | 1 | 1
Lymphocyte percentage decreased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 10 | 10
White blood cell count decreased (Investigations) | 9 | 10
Protein urine present (Investigations) | 0 | 1
Lymphocyte percentage increased (Investigations) | 2 | 2
Blood potassium decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Basophil percentage decreased (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 2
Lipids abnormal (Investigations) | 1 | 2
Monocyte percentage increased (Investigations) | 1 | 2
Bilirubin conjugated increased (Investigations) | 1 | 1
Eosinophil percentage decreased (Investigations) | 1 | 1
Protein total decreased (Investigations) | 0 | 8
Blood albumin decreased (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Frequent bowel movement (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
High density lipoprotein decreased (Investigations) | 0 | 1
Reticulocyte count increased (Investigations) | 0 | 1
Neutrophil percentage decreased (Investigations) | 3 | 4
Neutrophil percentage increased (Investigations) | 0 | 1
Tri-iodothyronine free decreased (Investigations) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other